CLINICAL TRIAL: NCT07090525
Title: Bevacizumab Combined With Cisplatin Versus Cisplatin Monotherapy in Malignant Serous Effusions-A Prospective Randomized Controlled Study
Brief Title: Bevacizumab Combined With Cisplatin Versus Cisplatin Monotherapy in Malignant Serous Effusions
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, director, Qingdao Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY202508203
Record Dates: First submitted 2025-07-16; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Overall Response Rate
Keywords: Bevacizumab; malignant serous effusions; Randomized study
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bevacizumab plus cisplatin arm (Experimental)
  Interventions: Drug: Intracavity injection of bevacizumab 7.5mg/kg plus cisplatin 40mg/m2
- cisplatin arm (Active Comparator): cisplatin 40mg/m2 intracavity injection
  Interventions: Drug: cisplatin 40mg/m2 intracavity injection

INTERVENTIONS:
Drug: Intracavity injection of bevacizumab 7.5mg/kg plus cisplatin 40mg/m2 — Intracavity injection of bevacizumab 7.5mg/kg plus cisplatin 40mg/m2, repeat use on 21st day if the serous effusion not controlled
  Arms: bevacizumab plus cisplatin arm
Drug: cisplatin 40mg/m2 intracavity injection — cisplatin 40mg/m2 intracavity injection
  Arms: cisplatin arm

SUMMARY:
The purpose of this study is to explore the efficacy and safety ofof bevacizumab plus cisplatin compare with cisplatin in the treatment of malignant serous effusion in patients with advanced adenocarcinoma

DETAILED DESCRIPTION:
This study is a prospective, three-center, randomized, phase II clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent;
2. Treatment naive serous effusion of patients with adenocarcinoma without activating gene mutation.
3. Eastern Cooperative Oncology Group (ECOG) score ≤ 2;
4. Survival is expected to exceed 3 months

Exclusion Criteria:

* The subject had received anti-vascular endothelial growth factor (VEGF) small molecule tyrosine kinase inhibitors or monoclonal antibodies in the past 4 weeks; The subject had participated any clinical trials in the past 4 weeks; The subject had previously received bevacizumab of pleural perfusion therapy;

Laboratory results:

White blood cell count <3 × 109 / L, neutrophil count <1.5 × 109 / L, platelet <75 × 109 / L, or hemoglobin <8g / dL; Coagulation abnormalities (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time (APTT) > 1.5 ULN), with bleeding tendency or being treated with thrombolysis or anticoagulation; Serum total bilirubin ≥1.5 ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 ULN in the absence of liver metastases; ALT or AST ≥5 ULN in liver metastases; Serum albumin <30g / L; Serum creatinine ≥ 1.5 ULN or creatinine clearance <40ml / min; Urine routine urinary protein ≥ ++, or 24 hours urine protein ≥ 1.0 g; Hypertension cannot be controlled by drugs; Heart disease with significant clinical symptoms, such as: congestive heart failure, coronary heart disease with symptom, arrhythmia hardly be controlled by drugs, myocardial infarction in 6 months, or heart failure; Imaging (CT or MRI) showed a tumor lesion 5 mm away from the large vessels, or the presence of invasive central vasculature of the central tumor; imaging (CT or MRI) showed significant cavitation or necrosis of the lung tumor; Other diseases that may cause haemoptysis; Imaging (CT or chest radiograph) showed significant pneumothorax, fluid pneumothorax; Bilateral pleural cavity to a large number of effusion or encapsulated pleural effusion; Obvious cough blood in 6 months, or daily hemoptysis amounted to half a teaspoon (2.5ml) or more; Significant bleeding symptoms or with definite bleeding tendency within 12 months before randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, occult blood ++ and above, intracerebral hemorrhage, vasculitis, or with congenital or acquired coagulopathy disorders; Thrombosis, cancer thrombosis (including arteriovenous thrombosis, tumor thrombus, pulmonary embolism, transient ischemic attack, etc.) occurred within 12 months; There are gastrointestinal obstruction, peptic ulcer, Crohn's disease, ulcerative colitis and other gastrointestinal diseases or other diseases may cause gastrointestinal bleeding or perforation; Severe respiratory diseases, or need long-term oxygen, corticosteroid treatment of diseases such as chronic obstructive pulmonary disease, interstitial lung disease and respiratory failure; The toxicity of previous antineoplastic therapies has not yet recovered to below grade 2 or has not fully recovered; Patients with uncontrolled central nervous system metastasis; There are serious uncontrolled systemic diseases, such as nephrotic syndrome, infection, poorly controlled diabetes; Patients with active HIV（human immunodeficiency virus）, HBV（hepatitis B virus）, or HCV（hepatitis C virus） infection; Patients had undergone surgery (<28 days) or did not heal completely, or had other unhealed wounds before the study; Patients known to be allergic to bevacizumab or any of the components of the drug; Pregnant or lactating female patients, or unwilling to take contraceptive measures of reproductive age patients (including men); There is a serious psychological or mental abnormality, or lack of compliance; The investigator determines other circumstances that may affect the conduct of clinical studies and the determination of findings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
overall response | 4 weeks
overall response | serous effusion ORR at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code